CLINICAL TRIAL: NCT01853033
Title: A Study in Patients With Rheumatoid Arthritis to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of ABT-122
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Subcutaneous Injections of ABT-122 in Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M14-048
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Tolerability; Immunogenicity; Safety; Rheumatoid Arthritis; Pharmacokinetics
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ABT-122

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Randomized 6 drug/2 placebo by group
  Interventions: Biological: ABT-122; Biological: Placebo
- Group 2 (Experimental): Randomized 6 drug/2 placebo by group
  Interventions: Biological: ABT-122; Biological: Placebo
- Group 3 (Experimental): Randomized 6 drug/2 placebo by group
  Interventions: Biological: ABT-122; Biological: Placebo

INTERVENTIONS:
Biological: ABT-122 — Injection
Biological: Placebo — Placebo Injection

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of ABT-122 in subjects with Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, multiple ascending dose study. Twenty-four subjects with Rheumatoid Arthritis will be selected to participate. Subjects will be randomized to receive either ABT-122 or placebo. ABT-122 or placebo will be administered as subcutaneous (under the skin) injections in three dosing groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis (RA) > 3 months.
* On methotrexate (MTX) therapy => 3 months and on a stable dose for at least 4 weeks.
* Except for MTX, must have discontinued all disease-modifying antirheumatic drugs (DMARDs) for at least 3 months or 5 half-lives, whichever is longer.
* Body Mass Index (BMI) is 19 to 38, inclusive.
* Other than RA, subjects should be in good general health.

Exclusion Criteria:

* Evidence of anti-ABT-122 antibody on a serum sample taken at Screening.
* History of significant allergic reaction; or history of anaphylactic reaction to any agent; or history of major reaction to any IgG containing product.
* History of persistent chronic or active infection(s) requiring hospitalization or treatment with intravenous or oral anti-microbials/antibiotics within the past 30 days.
* History or evidence of active tuberculosis (TB) or the subject has evidence of risk factor for latent TB.
* Subject has any medical condition or illness other than RA that is not well controlled with treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | From date of first dose of ABT-122 until 42 days after the last dose of ABT-122
  Collect all adverse events at each visit
Change in physical exam including vital signs | From date of first dose of ABT-122 until 42 days after last dose of ABT-122
  Blood pressure, pulse and body temperature
Change in clinical lab test results | From date of first dose of ABT-122 until 42 days after the last dose of ABT-122
  Hematology, Chemistry, and Urinalysis
Change in Electrocardiogram (ECG) results | From subject's baseline (prior to subject's first dose) and up to 168 hours following the last dose of study drug
  ECGs done in triplicate
Determination of pharmacokinetic (PK) parameters | Prior to first dose up to 42 days after the last dose of ABT-122
  Cmax, Tmax, AUC, elimination rate constant and half-life

SECONDARY OUTCOMES:
Measurement of anti-drug anti-bodies (ADA) of ABT-122 | Prior to each dose and up until 42 days after the last dose of ABT-122
  Measurement of ADA

CONTACTS AND LOCATIONS:
Overall Officials: Robert Padley, MD, Study Director — AbbVie
Locations (4):
- United States (4):
  - Site Reference ID/Investigator# 108655, Lenexa, Kansas
  - Site Reference ID/Investigator# 107115, Raleigh, North Carolina
  - Site Reference ID/Investigator# 118964, Duncansville, Pennsylvania
  - Site Reference ID/Investigator# 100780, Dallas, Texas

REFERENCES:
- [Result] Khatri A, Goss S, Jiang P, Mansikka H, Othman AA. Pharmacokinetics of ABT-122, a TNF-alpha- and IL-17A-Targeted Dual-Variable Domain Immunoglobulin, in Healthy Subjects and Patients with Rheumatoid Arthritis: Results from Three Phase I Trials. Clin Pharmacokinet. 2018 May;57(5):613-623. doi: 10.1007/s40262-017-0580-y. PMID 28744796
- [Derived] Fleischmann RM, Wagner F, Kivitz AJ, Mansikka HT, Khan N, Othman AA, Khatri A, Hong F, Jiang P, Ruzek M, Padley RJ. Safety, Tolerability, and Pharmacodynamics of ABT-122, a Tumor Necrosis Factor- and Interleukin-17-Targeted Dual Variable Domain Immunoglobulin, in Patients With Rheumatoid Arthritis. Arthritis Rheumatol. 2017 Dec;69(12):2283-2291. doi: 10.1002/art.40319. Epub 2017 Nov 8. PMID 28941216